CLINICAL TRIAL: NCT03025542
Title: A Multicenter, Randomized, Subject-Blind, Investigator-Blind Study to Evaluate the Time Course of Pharmacodynamic Response, Safety and Pharmacokinetics of Bimekizumab in Adult Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: A Study to Evaluate the Pharmacokinetics (PK), Pharmacodynamics (PD), and Safety of Bimekizumab in Patients With Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PS0016; 2016-002368-15 (EudraCT Number)
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Results first posted 2021-01-06 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-09

CONDITIONS: Chronic Plaque Psoriasis
Keywords: Psoriasis; Chronic Plaque Psoriasis; Bimekizumab
MeSH Terms: conditions — Psoriasis | interventions — bimekizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is an Investigator- and Subject-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm 1 (Experimental): Subjects randomized in this arm will receive a combination of Bimekizumab and Placebo injections.
  Interventions: Drug: Bimekizumab; Other: Placebo
- Treatment Arm 2 (Experimental): Subjects randomized in this arm will receive Bimekizumab injections.
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Based on their randomization subjects will receive a combination of several injections of Bimekizumab.
  Other Names: UCB4940
Other: Placebo — Subjects will receive injections of Placebo.
  Arms: Treatment Arm 1

SUMMARY:
This is a Phase 2a, multicenter, randomized, subject-blind, investigator-blind, study to investigate the pharmacokinetics (PK), pharmacodynamics (PD), and safety of bimekizumab in adult subjects with moderate to severe chronic plaque psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age and less than or equal to 70
* Chronic plaque psoriasis for at least 6 months prior to Screening
* Psoriasis Area and Severity Index (PASI) >=12 and body surface area (BSA) >=10% and Investigator's Global Assessment (IGA) score >=3 on a 5-point scale
* Candidates for systemic psoriasis therapy and/or phototherapy and/or chemophototherapy
* Female subjects must be postmenopausal, permanently sterilized or, if of childbearing potential, must be willing to use a highly effective method of contraception up till 20 weeks after last administration of study drug, and have a negative pregnancy test at Visit 1 (Screening) and immediately prior to first dose
* Male subjects with a partner of childbearing potential must be willing to use a condom when sexually active, up till 20 weeks after the last administration of study medication (anticipated 5 half-lives)

Exclusion Criteria:

* Subjects previously participating in a bimekizumab study
* Subjects with erythrodermic, guttate, pustular form of psoriasis, or drug-induced psoriasis
* History of chronic or recurrent infections, or a serious or life-threatening infection within the 6 months prior to the Baseline Visit (including herpes zoster)
* High risk of infection in the Investigator's opinion
* Current sign or symptom that may indicate an active infection
* Concurrent acute or chronic viral hepatitis B or C or human immunodeficiency virus (HIV) infection
* Live (includes attenuated) vaccination within the 8 weeks prior to Baseline
* Subjects with concurrent malignancy or history of malignancy during the past 5 years (except for specific malignant condition as defined in the protocol)
* Primary immunosuppressive conditions
* TB infection, high risk of acquiring TB infection, latent TB infection (LTBI), or current or history of NTMB infection
* Laboratory abnormalities, as defined in the study protocol
* Any condition which, in the Investigator's judgement, would make the subject unsuitable for inclusion in the study
* Exposure to more than 1 biological response modifier (limited to anti-TNF or IL-12/-23) or any biologic response modifier during the three months prior to the Baseline Visit
* Subjects have received previous treatment with any anti-IL-17 therapy for the treatment of psoriasis or psoriatic arthritis
* Subjects with a diagnosis of inflammatory conditions other than psoriasis or psoriatic arthritis, including but not limited to rheumatoid arthritis, sarcoidosis, or systemic lupus erythematosus. Subjects with a diagnosis of Crohn's disease or ulcerative colitis are allowed as long as they have no active symptomatic disease at Screening or Baseline
* Subjects taking psoriatic arthritis medications other than nonsteroidal anti-inflammatory drugs (NSAIDs) or analgesics

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273(UCB)
Locations (8):
- Ps0016 704, Bexley, Ohio, United States
- Australia (3):
  - Ps0016 102, Kogarah
  - Ps0016 101, Melbourne
  - Ps0016 104, Woolloongabba
- Canada (3):
  - Ps0016 201, Ajax
  - Ps0016 203, London
  - Ps0016 202, Windsor
- Ps0016 501, Chisinau, Moldova

REFERENCES:
- [Result] Oliver R, Krueger JG, Glatt S, Vajjah P, Mistry C, Page M, Edwards H, Garcet S, Li X, Dizier B, Maroof A, Watling M, El Baghdady A, Baeten D, Ionescu L, Shaw S. Bimekizumab for the treatment of moderate-to-severe plaque psoriasis: efficacy, safety, pharmacokinetics, pharmacodynamics and transcriptomics from a phase IIa, randomized, double-blind multicentre study. Br J Dermatol. 2022 Apr;186(4):652-663. doi: 10.1111/bjd.20827. Epub 2021 Dec 27. PMID 34687214
- [Result] Gordon KB, Langley RG, Warren RB, Okubo Y, Stein Gold L, Merola JF, Peterson L, Wixted K, Cross N, Deherder D, Thaci D. Bimekizumab Safety in Patients With Moderate to Severe Plaque Psoriasis: Pooled Results From Phase 2 and Phase 3 Randomized Clinical Trials. JAMA Dermatol. 2022 Jul 1;158(7):735-744. doi: 10.1001/jamadermatol.2022.1185. PMID 35544084
- See also: Product Information — https://www.ema.europa.eu/en/documents/product-information/bimzelx-epar-product-information_en.pdf
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in December 2016 and concluded in December 2017.
Pre-assignment Details: Participant Flow refers to the Safety Set (SS).
Groups:
- Bimekizumab 320 mg + PBO: Bimekizumab 320 milligrams (mg) administered subcutaneously (sc) at Baseline and Week 4, and placebo administered at Week 16.
- Bimekizumab 320 mg: Bimekizumab 320 mg administered sc at Baseline and Weeks 4 and 16.
Period: Overall Study
Arm/Group | Bimekizumab 320 mg + PBO | Bimekizumab 320 mg
Started | 32 | 17
Completed | 30 | 15
Not Completed | 2 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set (SS) which consisted of all participants who received at least 1 dose of the study medication.
Arm/Group | Bimekizumab 320 mg + PBO | Bimekizumab 320 mg | Total Title
Number analyzed (Participants) | 32 | 17 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 16 | 46
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (14.1) | 45.9 (10.4) | 43.2 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 6 | 23
  Male | 15 | 11 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 4 | 5
  Black or African American | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 30 | 12 | 42

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) at Week 28
Description: The PASI is the most commonly used and validated assessment for grading the severity of psoriasis in clinical studies. The PASI quantifies the severity and extent of the disease and weighs these with the percentage of body surface area (BSA) involvement. The percent area of involvement (BSA%) is estimated across 4 body areas; head (10%), upper limbs (20%), trunk (30%), and lower limbs (40%) and then transferred into a grade. The Investigator assesses the average redness, thickness, and scaliness of lesions in each body area (each on a 5 point scale); 0=none, 1=slight, 2=moderate, 3=marked, and 4=very marked. The PASI score ranges from 0 to 72 with a higher score indicating increased disease severity.
Time Frame: From Baseline to Week 28
Population: The Full Analysis Set (FAS) consisted of all randomized participants who received at least 1 dose of the study medication and have a valid measurement of the primary efficacy variable post Baseline.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Bimekizumab 320 mg + PBO (FAS): Bimekizumab 320 mg administered subcutaneously (sc) at Baseline and Week 4, and placebo administered at Week 16. Participants formed the Full Analysis Set (FAS).
- Bimekizumab 320 mg (FAS): Bimekizumab 320 mg administered sc at Baseline and Weeks 4 and 16. Participants formed the Full Analysis Set (FAS).
Arm/Group | Bimekizumab 320 mg + PBO (FAS) | Bimekizumab 320 mg (FAS)
Number analyzed (Participants) | 32 | 17
scores on a scale | -10.76 (7.58) | -19.74 (8.77)

2. Primary Outcome: Plasma Concentration of Bimekizumab at Baseline
Description: Plasma concentration was expressed as geometric mean concentrations (GMCs) and measured in micrograms per milliliter (μg/mL). Note: Means, Lower confidence interval (LCI), Upper confidence interval (UCI) are only calculated if at least 2/3 of the concentrations were quantified at the respective time point. Values below limit of quantification (BLQ) are replaced by value of lower limit of quantification (LLOQ)/2 (=0.075ug/mL) in calculations of means.
Time Frame: at Baseline
Population: The Pharmacokinetics Per-Protocol Set (PK-PPS) consisted of all randomized participants who received at least 1 dose of the study medication and provided at least 1 quantifiable plasma concentration post-dose. Number of participants analyzed reflects Baseline.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Groups:
- Bimekizumab 320 mg + PBO (PK-PPS): Bimekizumab 320 mg administered subcutaneously (sc) at Baseline and Week 4, and placebo administered at Week 16. Participants formed the Pharmacokinetics Per-Protocol Set (PK-PPS).
- Bimekizumab 320 mg (PK-PPS): Bimekizumab 320 mg administered sc at Baseline and Weeks 4 and 16. Participants formed the Pharmacokinetics Per-Protocol Set (PK-PPS).
Arm/Group | Bimekizumab 320 mg + PBO (PK-PPS) | Bimekizumab 320 mg (PK-PPS)
Number analyzed (Participants) | 32 | 17
μg/mL | NA [NA to NA] — Values were below the level of detection; Participants had no prior BKZ treatment. | NA [NA to NA] — Values were below the level of detection; Participants had no prior BKZ treatment.

3. Primary Outcome: Plasma Concentration of Bimekizumab at Week 2
Description: as for outcome 2
Time Frame: at Week 2
Population: The Pharmacokinetics Per-Protocol Set (PK-PPS) consisted of all randomized participants who received at least 1 dose of the study medication and provided at least 1 quantifiable plasma concentration post-dose. Number of participants analyzed reflects Week 2.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Bimekizumab 320 mg + PBO (PK-PPS) | Bimekizumab 320 mg (PK-PPS)
Number analyzed (Participants) | 32 | 16
μg/mL | 19.749 [17.0 to 23.0] | 14.437 [10.8 to 19.3]

4. Primary Outcome: Plasma Concentration of Bimekizumab at Week 4
Description: as for outcome 2
Time Frame: at Week 4
Population: The Pharmacokinetics Per-Protocol Set (PK-PPS) consisted of all randomized participants who received at least 1 dose of the study medication and provided at least 1 quantifiable plasma concentration post-dose. Number of participants analyzed reflects Week 4.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Bimekizumab 320 mg + PBO (PK-PPS) | Bimekizumab 320 mg (PK-PPS)
Number analyzed (Participants) | 31 | 17
μg/mL | 11.402 [9.7 to 13.4] | 9.077 [7.2 to 11.5]

5. Primary Outcome: Plasma Concentration of Bimekizumab at Week 8
Description: as for outcome 2
Time Frame: at Week 8
Population: The Pharmacokinetics Per-Protocol Set (PK-PPS) consisted of all randomized participants who received at least 1 dose of the study medication and provided at least 1 quantifiable plasma concentration post-dose. Number of participants analyzed reflects Week 8.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Bimekizumab 320 mg + PBO (PK-PPS) | Bimekizumab 320 mg (PK-PPS)
Number analyzed (Participants) | 31 | 16
μg/mL | 16.728 [14.4 to 19.5] | 13.969 [11.1 to 17.6]

6. Primary Outcome: Plasma Concentration of Bimekizumab at Week 12
Description: as for outcome 2
Time Frame: at Week 12
Population: The Pharmacokinetics Per-Protocol Set (PK-PPS) consisted of all randomized participants who received at least 1 dose of the study medication and provided at least 1 quantifiable plasma concentration post-dose. Number of participants analyzed reflects Week 12.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Bimekizumab 320 mg + PBO (PK-PPS) | Bimekizumab 320 mg (PK-PPS)
Number analyzed (Participants) | 31 | 15
μg/mL | 5.972 [4.9 to 7.3] | 5.466 [3.9 to 7.7]

7. Primary Outcome: Plasma Concentration of Bimekizumab at Week 16
Description: Plasma concentration was expressed as geometric mean concentrations (GMCs) and measured in micrograms per milliliter (µg/mL). Note: Means, Lower confidence interval (LCI), Upper confidence interval (UCI) are only calculated if at least 2/3 of the concentrations were quantified at the respective time point. Values below limit of quantification (BLQ) are replaced by value of lower limit of quantification (LLOQ)/2 (=0.075ug/mL) in calculations of means.
Time Frame: at Week 16
Population: The Pharmacokinetics Per-Protocol Set (PK-PPS) consisted of all randomized participants who received at least 1 dose of the study medication and provided at least 1 quantifiable plasma concentration post-dose. Number of participants analyzed reflects Week 16.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Bimekizumab 320 mg + PBO (PK-PPS) | Bimekizumab 320 mg (PK-PPS)
Number analyzed (Participants) | 31 | 15
µg/mL | 2.200 [1.6 to 3.0] | 2.293 [1.4 to 3.7]

8. Primary Outcome: Plasma Concentration of Bimekizumab at Week 20
Description: as for outcome 2
Time Frame: at Week 20
Population: The Pharmacokinetics Per-Protocol Set (PK-PPS) consisted of all randomized participants who received at least 1 dose of the study medication and provided at least 1 quantifiable plasma concentration post-dose. Number of participants analyzed reflects Week 20.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Bimekizumab 320 mg + PBO (PK-PPS) | Bimekizumab 320 mg (PK-PPS)
Number analyzed (Participants) | 31 | 15
μg/mL | 0.798 [0.5 to 1.2] | 9.702 [7.3 to 13.0]

9. Primary Outcome: Plasma Concentration of Bimekizumab at Week 24
Description: as for outcome 2
Time Frame: at Week 24
Population: The Pharmacokinetics Per-Protocol Set (PK-PPS) consisted of all randomized participants who received at least 1 dose of the study medication and provided at least 1 quantifiable plasma concentration post-dose. Number of participants analyzed reflects Week 24.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Bimekizumab 320 mg + PBO (PK-PPS) | Bimekizumab 320 mg (PK-PPS)
Number analyzed (Participants) | 29 | 15
μg/mL | NA [NA to NA] — Values were below the level of detection. | 4.377 [3.2 to 6.0]

10. Primary Outcome: Plasma Concentration of Bimekizumab at Week 28
Description: as for outcome 2
Time Frame: at Week 28
Population: The Pharmacokinetics Per-Protocol Set (PK-PPS) consisted of all randomized participants who received at least 1 dose of the study medication and provided at least 1 quantifiable plasma concentration post-dose. Number of participants analyzed reflects Week 28.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Bimekizumab 320 mg + PBO (PK-PPS) | Bimekizumab 320 mg (PK-PPS)
Number analyzed (Participants) | 26 | 13
μg/mL | NA [NA to NA] — Values were below the level of detection. | 1.933 [1.2 to 3.1]

11. Primary Outcome: Plasma Concentration of Bimekizumab at Week 36
Description: as for outcome 2
Time Frame: at Week 36
Population: The Pharmacokinetics Per-Protocol Set (PK-PPS) consisted of all randomized participants who received at least 1 dose of the study medication and provided at least 1 quantifiable plasma concentration post-dose. Number of participants analyzed reflects Week 36.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Bimekizumab 320 mg + PBO (PK-PPS) | Bimekizumab 320 mg (PK-PPS)
Number analyzed (Participants) | 24 | 14
μg/mL | NA [NA to NA] — Values were below the level of detection. | 0.322 [0.2 to 0.6]

12. Primary Outcome: Percentage of Participants Reporting Positive Anti-Drug-Antibodies (ADA) Titre Prior to Study Treatment With Bimekizumab at Baseline
Description: An ADA status of positive was concluded for any participant with an ADA level that was above cut point (ACP) and 'confirmed positive' (CP) at any time point. A participant was classified as having treatment-induced ADA positivity when meeting one of the following criteria: -The Baseline result was either below cut point (BCP) or ACP and 'not confirmed positive' (NCP), and at least 1 post Baseline time point was ACP and CP. -The Baseline result was positive (ACP and CP) and at least one post-Baseline measurement showed a pre-defined fold increase in titre from the Baseline value. Note: The overall status of a participant is 'Positive' if at any post-Baseline visit the result was ACP and confirmed positive.
Time Frame: at Baseline
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the study medication. Percentages were based on the number of participants with a non-missing measurement at Baseline.
Measure: Number; unit: percentage of participants
Groups:
- Bimekizumab 320 mg + PBO (SS): Bimekizumab 320 mg administered subcutaneously (sc) at Baseline and Week 4, and placebo administered at Week 16. Participants formed the Safety Set (SS).
- Bimekizumab 320 mg (SS): Bimekizumab 320 mg administered sc at Baseline and Weeks 4 and 16. Participants formed the Safety Set (SS).
Arm/Group | Bimekizumab 320 mg + PBO (SS) | Bimekizumab 320 mg (SS)
Number analyzed (Participants) | 32 | 17
percentage of participants | 3.1 | 0

13. Primary Outcome: Percentage of Participants Reporting an Overall Positive Anti-Drug-Antibodies (ADA) Titre Following Study Treatment With Bimekizumab
Description: as for outcome 12
Time Frame: From Baseline to Safety Follow-Up Visit (Week 36)
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 320 mg + PBO (SS) | Bimekizumab 320 mg (SS)
Number analyzed (Participants) | 32 | 17
percentage of participants | 34.4 | 47.1

14. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Events (AEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. Within the Safety Set, this trial reported a total of 164 occurences of adverse events, of which 7 were pre-treatment adverse events and 157 were treatment-emergent adverse events (TEAEs).
Time Frame: From Screening to Safety Follow-Up Visit (Week 36)
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 320 mg + PBO (SS) | Bimekizumab 320 mg (SS)
Number analyzed (Participants) | 32 | 17
percentage of participants | 87.5 | 88.2

15. Secondary Outcome: Percentage of Participants Achieving a 75% or Higher Improvement From Baseline in PASI (Psoriasis Area and Severity Index) Score at Week 16
Description: The PASI75 response assessments are based on at least 75% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: From Baseline to Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 320 mg + PBO (FAS) | Bimekizumab 320 mg (FAS)
Number analyzed (Participants) | 32 | 17
percentage of participants | 93.8 | 88.2

16. Secondary Outcome: Percentage of Participants Achieving a 90% or Higher Improvement From Baseline in PASI (Psoriasis Area and Severity Index) Score at Week 16
Description: The PASI90 response assessments are based on at least 90% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: From Baseline to Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 320 mg + PBO (FAS) | Bimekizumab 320 mg (FAS)
Number analyzed (Participants) | 32 | 17
percentage of participants | 84.4 | 70.6

17. Secondary Outcome: Percentage of Participants Achieving a 100% Improvement From Baseline in PASI (Psoriasis Area and Severity Index) Score at Week 16
Description: The PASI100 response assessments are based on at least 100% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: From Baseline to Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 320 mg + PBO (FAS) | Bimekizumab 320 mg (FAS)
Number analyzed (Participants) | 32 | 17
percentage of participants | 46.9 | 52.9

18. Secondary Outcome: Percentage of Participants With IGA (Investigator´s Global Assessment) Response at Week 16
Description: The Investigator's Global Assessment (IGA) measures the overall psoriasis severity following a 5-point scale (0-4), where scale 0= clear, no signs of psoriasis; presence of post-inflammatory hyperpigmentation, scale 1= almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2= mild thickening, pink to light red coloration and predominately fine scaling, 3= moderate, clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling and 4= severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions.
Time Frame: at Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 320 mg + PBO (FAS) | Bimekizumab 320 mg (FAS)
Number analyzed (Participants) | 32 | 17
percentage of participants | 81.3 | 64.7

ADVERSE EVENTS:
Time Frame: From Baseline to Week 36
Arm/Group | Bimekizumab 320 mg + PBO (SS) | Bimekizumab 320 mg (SS)
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/17
Serious Adverse Events (participants affected / at risk) | 2/32 | 1/17
Other Adverse Events (participants affected / at risk) | 28/32 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bimekizumab 320 mg + PBO (SS) (N=32) | Bimekizumab 320 mg (SS) (N=17)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bimekizumab 320 mg + PBO (SS) (N=32) | Bimekizumab 320 mg (SS) (N=17)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-alcoholic fatty liver (Hepatobiliary disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 6 (8) | 3 (3)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (3)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 1 (1)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 2 (2)
Bacterial diarrhoea (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 2 (4) | 3 (7)
White blood cell count decreased (Metabolism and nutrition disorders) | 2 (2) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (4)
Neutrophil count decreased (Investigations) | 1 (1) | 3 (3)
Blood cholesterol increased (Investigations) | 1 (1) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Mean cell haemoglobin concentration decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (6) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-09-23): https://cdn.clinicaltrials.gov/large-docs/42/NCT03025542/Prot_002.pdf
  • Statistical Analysis Plan (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT03025542/SAP_003.pdf